CLINICAL TRIAL: NCT05171998
Title: Characterisation of the Immune Response to SARS-CoV-2 and Other Common Infections in Type 1 Diabetes
Brief Title: Characterisation of the Immune Response to SARS-CoV-2 Infection / COVID-19 in Type 1 Diabetes
Acronym: TIRID
Status: Completed | Type: Observational
Sponsor: Cwm Taf University Health Board (NHS) (Other Government)
Collaborators: Cardiff University (Other); University of Oxford (Other); Imperial College London (Other)
Responsible Party: Sponsor
Other Study IDs: CT 253888
Record Dates: First submitted 2021-12-23; First posted 2021-12-29 (Actual); Last update posted 2024-08-15 (Actual); Status verified 2024-03

CONDITIONS: SARS-CoV2 Infection Common Pathogens; Diabetes Mellitus, Type 1
MeSH Terms: conditions — Diabetes Mellitus, Type 1 | interventions — Hematologic Tests

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — whole venous blood including peripheral blood mononuclear cells and serum.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Procedure: venous blood sample — Phlebotomy procedure for a venous blood draw.
  Other Names: blood tests

SUMMARY:
Emerging clinical details of the current SARS-CoV-2 pandemic have illustrated that there are multiple clinical presentations and outcomes of this viral infection. People with an infection have been reported to have a spectrum of disease from severe acute respiratory distress requiring ventilation, to mild respiratory or gastrointestinal symptoms and asymptomatic presentations. The SARS-CoV-2 pandemic has been accompanied with a substantial increase in the number of individuals presenting with new onset type 1 diabetes [1]. Most individuals presenting with type 1 diabetes since the start of the COVID-19 pandemic are SARS-CoV-2 antibody positive. These findings suggest that SARS-CoV-2 infection can cause type 1 diabetes. Investigators have identified that many individuals presenting with type 1 diabetes since the start of the COVID-19 pandemic are SARS-CoV-2 positive by swab or blood test. Researchers have also observed that T cells in patients who have had COVID recognise some of the peptides in the pancreatic islet cells, which are responsible for production of insulin. These findings suggest that SARS-CoV-2 infection may be associated with new onset of type 1 diabetes.

The aim of this project is to understand the host immune response to infection with SARS-CoV-2 and other common pathogens over time in convalescent newly diagnosed patients with type 1 diabetes, including acquired immune responses, gene expression profiling in peripheral blood and to identify host genetic variants associated with disease progressions or severity. Participants will have Type 1 diabetes and will have had a diagnosis of COVID-19 (confirmed by a positive nasopharyngeal swab PCR test and/or SARS-CoV-2 antibody test) and have recovered from COVID-19. Samples will be processed and analysed to explore the molecular mechanisms by which SARS-CoV-2 and other common infections might precipitate immune attack on insulin-producing cells resulting in autoimmune diabetes.

DETAILED DESCRIPTION:
AIMS AND OBJECTIVES The objective of this project is to understand the host immune response to infection with SARS-CoV-2 and other common infections over time in convalescent patients that develop type 1 diabetes (T1D). Preliminary data show that diabetogenic T-cells in patients that developed T1D before 2019 can recognise SARS-CoV-2 and other common human pathogens. If the reverse is true, it would provide a plausible mechanism for the development of T1D following SARS-CoV-2 or some common infections. We would like to ascertain why some people develop T1D after infection.

Primary objectives are to determine whether individuals that develop T1D following infection bear the HLA A*0201 and HLA*2402 genes known to be associated with T1D and to show that SARS-CoV-2/pathogen-specific killer T-cells in these individuals are capable of directly destroying insulin-producing pancreatic beta cells. The ability of pathogen-specific T-cells to recognise diabetogenic T-cell epitopes will be examined using peptide-HLA multimers. Cross-reactive T-cell receptors will be manufactured for biophysical and structural analyses to enable an understanding of how SARS-CoV-2 and other common infectious agents might induce T1D.

Methodology will examine whether convalescent patients that develop T1D predominantly express the human leukocyte antigens (HLAs) HLA A*02 and HLA*24 by staining a small part of the sample with antibodies for these HLA. Investigators anticipate that there could be a large enrichment for these disease risk HLA (>75% of patients expressing one of these disease-risk alleles) [2]. T-cell library [3] and peptide-HLA multimer [4-6] approaches will be used to isolate T-cells that recognise epitopes from SARS-CoV-2 and other common pathogens via HLA A*02 and HLA*24. The monoclonal T-cell populations generated will be tested for recognition of known diabetogenic epitopes present on the surface of human pancreatic beta cells. Where such T-cell cross-reactivity [7] is identified the team will sequence the complementarity determining region of the cognate T-cell receptor so that it can be manufactured as a soluble protein [8] for further biophysical and structural studies [9,10] aimed at understanding how SARS-CoV-2 and other common pathogens might induce T1D in a minority of individuals.

The study will be prospective, observational study. Participants will be convalescent patients with recent new diagnosis of type 1 diabetes (n=30). Eligible participants will be identified and referred from Consultant Paediatric Endocrinologists at The Department of Child Health at Cwm Taf Morgannwg University Health board, The Department of Child Health, Cardiff and the Vale health board and Department of Child Health, St, Mary's Hospital, London who are all part of the clinical research study team and direct clinical care team. All participants and their parents /guardians will receive a participant information sheet and have time and privacy to read and understand the content. A member of the study team trained in Good Clinical Practice will be available to provide support and answer any questions. Informed consent will then be gained in writing on a consent form, or in the case of paediatric participants on an assent form and a Parent/Guardian consent form. Participants will be issued with a unique study number.

A sample of blood will be taken by a trained phlebotomist, 50mls (or less in children according to the participant's weight). The sample will be anonymised and issued with the unique study number. We will require peripheral blood mononuclear cells (PBMC) from of blood on the day of recruitment. Anonymised blood samples will be transferred for T cell research and Cwm Taf University Health board laboratory for serology tests (Roche SARS-CoV-2 IgM and IgG assay at a UKAS accredited laboratory) with appropriate UN3373 packaging. Samples will be used for immunological, virological and host genetic assays. Bloods will be processed to isolate serum and PBMC, including host RNA and DNA. T-cell libraries will be established using the PBMC. T-cell clones generated will be tested for cross-reactivity with established diabetogenic T-cell epitopes. The T-cell receptors (TCRs) will be manufactured from cross-reactive T-cells for further study. PBMC samples will also be stained with cognate peptide-HLA multimers using flow cytometry. This will generate information about their phenotype and activation status.

A Lay Description:

The blood will be separated into constituent parts using a thick density gradient solution and a centrifuge. The white blood cell layer, or PBMCs, is isolated from other parts of the blood and retained. All other parts are discarded in a bleach solution PBMCs are further processed to isolate the T-cells, these cells can then go down one of five routes:

1. The cells are treated to extract the DNA/RNA, and the DNA/RNA is analysed to gain information about the T-cell receptors and other associated molecules. The cells are killed during DNA/RNA extraction.
2. The cells will undergo genetic editing to provide information about the processes involved in normal T-cell function. Cells will be cultured for 28 days post gene editing, will undergo multiple rounds of division, and become non-relevant in terms of the Human Tissue Authority (HTA) act 2004.
3. The cells will be used in an assay where they are exposed to overlapping bits of SARS-CoV-2 proteins, they will then be grown in culture for 14 days after which time the cells will have undergone division and will be no longer HTA relevant. Cells that respond to SARS-CoV-2 proteins will be tested to see whether they have capacity to destroy insulin-producing pancreatic beta cells.
4. Using an automated sorter and fluorescent markers, the cells are sorted and analysed. Cells will die during this process which takes place on the day cells are processed in the lab.
5. Cells will be used in plate-based assays to learn about the processes involved in T-cell functions. Cells will be disposed after the assay which can take between 1 and 3 days depending on type of assay used.

This methodology was designed following Patient and Public Involvement, which were conducted remotely due to social distancing.

ELIGIBILITY:
Inclusion Criteria:

* Participants must be 8 years or more old
* Participants must have the capacity to provide consent or assent after discussing the participant information sheet, with consent gained from their parent/guardian
* Diagnosis of Type 1 diabetes during the course of the COVID pandemic.

Exclusion Criteria:

Participants under 8 years old.

* Inability to provide consent or assent/parental consent

Ages: 8 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Patients diagnosed with new Type 1 diabetes.
Sampling Method: Non-Probability Sample
Enrollment: 30 (Actual)
Dates: Start 2021-01-01 (Actual); Primary Completion 2024-07-01 (Actual); Study Completion 2024-07-01 (Actual)

PRIMARY OUTCOMES:
To determine whether SARS-CoV-2-specific T-cells cross-react with insulin producing cells in the pancreas of people with Type 1 diabetes. | One blood draw at time of first diagnosis of Type 1 diabetes
  To measure if SARS-CoV-2-specific/infection-specific T-cells can cross-recognise insulin producing cells in the pancreas to potentially cause loss of insulin and type 1 diabetes.

SECONDARY OUTCOMES:
To determine if expression of HLA A*02 and/or HLA A*24 is more common in Type 1 diabetes patients with SARS-CoV-2 cross-reactive T cells | 6 months
  To determine if individuals that develop type 1 diabetes following SARS-CoV-2 and other common infections are enriched for expression of HLA A*02 and/or HLA A*24

CONTACTS AND LOCATIONS:
Overall Officials: Rhian Beynon, Study Director — Cwm Taf University Health Board (NHS)
Locations (1):
- Cwm Taf Morgannwg University Health board, Llantrisant, Rhondda Cynon Taf, United Kingdom

IPD SHARING:
Plan to Share IPD: No